CLINICAL TRIAL: NCT01670344
Title: Virtual Implant Planning System - A Method to Support Image-guided Surgical Interventions
Brief Title: Evaluation of an Innovative Medical Device Supporting Orthopedic Surgical Interventions
Acronym: VIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Healthcare QT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10308644 Final 2.5
Record Dates: First submitted 2012-08-15; First posted 2012-08-22 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Fracture of Distal End of Radius
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Treatment with investigational method (virtual implant positioning system)
  Interventions: Procedure: Treatment with investigational method (virtual implant positioning system)
- B (Other): Treatment with surgical standard of care
  Interventions: Procedure: Treatment with surgical standard of care

INTERVENTIONS:
Procedure: Treatment with investigational method (virtual implant positioning system)
  Arms: A
Procedure: Treatment with surgical standard of care
  Arms: B

SUMMARY:
This study is a randomized, controlled, 2-arm, open trial to evaluate an innovative positioning system in the clinical setting of orthopedic surgery.

Aim of the study is the validation and comparison of the innovative medical device with the current standard method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diastal fracture of the radius
* Patients with the mentioned fracture and indication for surgical treatment according to national guidelines
* Age >/= 18 years of age
* Patients willing to participate and after having given their informed consent in written form

Exclusion Criteria:

* Participation in other interventional clinical trials
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of screw replacements in both treatments arms | Participants will be followed for the duration of the hospital stay, an expected average of 3 days
  The number of screw replacements in both treatment arms will be assessed to evaluate the investigational method in comparison to the standard of care (arm B)

SECONDARY OUTCOMES:
Comparison of the investigational method to the standard of care regarding radiation time. | Participants will be followed for the duration of the hospital stay, an expected average of 3 days
Number of adverse events and serious adverse events during the clinical investigarion. | Participants will be followed for the duration of the hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Kleinszig Gerhard, MSc, Study Director — Sponsor GmbH
Locations (1):
- Siemens AG Healthcare Sector, Erlangen, Germany